CLINICAL TRIAL: NCT02625766
Title: Impact of Surgery on Pain in Lateral Compression Type Pelvic Fractures: a Prospective Trial
Brief Title: Pelvis RCT: Impact of Surgery on Pain in Lateral Compression Type Pelvic Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Robert O'Toole, Head of the UM SOM's Division of Orthpaedic Traumatology and Chief of Orthopaedics for the University of Maryland Medical Center's (UMMC) R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00060038
Record Dates: First submitted 2015-11-19; First posted 2015-12-09 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: LC Pelvic Fracture
Keywords: Operative vs. Non-operative; LC pelvic fracture; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operative (Experimental): Patients enrolled in the operative treatment group will undergo surgical intervention for their pelvic fracture. The surgeon will decide the best surgical technique as per standard of care for the patient's injury. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments to determine if the injury is healing properly. If additional surgery is required or other complications arise, this will be recorded within the study follow-up forms.
  Interventions: Procedure: LC fracture surgical fixation
- Non-operative (Experimental): Patients enrolled in the non-operative treatment group will not undergo surgical intervention for their pelvic fracture. They will mobilize as per the surgeon's instructions according to standard of care of for this injury. X-rays will be taken at follow-up clinic appointments to determine if the injury is healing properly or if the pelvis has shifted and may warrant surgical intervention. If complications arise and/or surgery is required, crossover will be allowed and recorded within study follow-up forms.
  Interventions: Procedure: LC fracture non-operative management

INTERVENTIONS:
Procedure: LC fracture surgical fixation
  Arms: Operative
Procedure: LC fracture non-operative management
  Arms: Non-operative

SUMMARY:
Lateral compression type pelvic ring injuries remain the most common type of pelvic fractures encountered. There is a substantial amount of controversy surrounding the treatment of these injuries and there is evidence that both operative and non-operative treatment can be successful.

DETAILED DESCRIPTION:
The crux of the problem is determining which of these patients would benefit from early surgical stabilization and which will heal uneventfully without surgery. Many authors site patient pain and inability to mobilize as indications for surgery, although there is conflicting evidence supporting this claim. The presence of chronic pain in the trauma population is a growing area of interest, and there is a push towards controlling pain more effectively in the acute setting. It remains to be proven that surgical intervention is more effective at decreasing acute and longer term pain.

There is evidence in the literature to support both operative and non-operative treatment of patients with LC1 or LC2 pelvic fractures. There is conflicting evidence that surgical stabilization decreases acute pain and narcotic requirements, although patients are often counseled to that effect. The investigators propose to prospectively randomize patients with lateral compression type pelvic fractures to non-operative versus operative treatment and track which group has less pain, less need for narcotic pain medications, and who mobilizes with physical therapy faster.

ELIGIBILITY:
Inclusion Criteria:

* The patient has one of the following pelvic fractures (includes bilateral sacral fractures): Lateral compression type 1, Lateral compression type 2, Lateral compression type 3
* The patient is between 18 and 80 years of age, inclusive
* The patient has reached skeletal maturity
* The patient's pelvic fracture is a result of trauma (includes polytraumatized patients)
* The patient/family/guardian is English-speaking
* The patient's surgeon agrees to randomization (the patient is amendable to either operative or non-operative treatment)
* Patient enrollment and, if applicable, patient randomization can occur within 96 hours post injury

Exclusion Criteria:

* The patient has prior surgical hardware in place that precludes intervention
* The patient's pelvic fracture is classified as a Lateral compression type 1 and the associated sacral fracture is incomplete as indicated by failure to violate both the anterior and posterior cortex
* The patient received prior surgical intervention for his/her current pelvic injury
* The patient has sacral morphology that precludes percutaneous fixation
* The patient is non-ambulatory due to an associated spinal cord injury
* The patient was non-ambulatory pre-injury
* The patient is currently pregnant
* The patient is enrolled in another research study that does not allow co-enrollment
* The patient is likely to have severe problems with maintaining follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O'Toole, MD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - Indiana University Health, Indianapolis, Indiana
  - University of Maryland, Shock Trauma Center, Baltimore, Maryland

REFERENCES:
- [Background] Young JW, Burgess AR, Brumback RJ, Poka A. Lateral compression fractures of the pelvis: the importance of plain radiographs in the diagnosis and surgical management. Skeletal Radiol. 1986;15(2):103-9. doi: 10.1007/BF00350202. PMID 3961516
- [Background] Manson T, O'Toole RV, Whitney A, Duggan B, Sciadini M, Nascone J. Young-Burgess classification of pelvic ring fractures: does it predict mortality, transfusion requirements, and non-orthopaedic injuries? J Orthop Trauma. 2010 Oct;24(10):603-9. doi: 10.1097/BOT.0b013e3181d3cb6b. PMID 20871246
- [Background] Lindahl J, Hirvensalo E. Outcome of operatively treated type-C injuries of the pelvic ring. Acta Orthop. 2005 Oct;76(5):667-78. doi: 10.1080/17453670510041754. PMID 16263614
- [Background] Routt ML Jr, Kregor PJ, Simonian PT, Mayo KA. Early results of percutaneous iliosacral screws placed with the patient in the supine position. J Orthop Trauma. 1995 Jun;9(3):207-14. doi: 10.1097/00005131-199506000-00005. PMID 7623172
- [Background] Bruce B, Reilly M, Sims S. OTA highlight paper predicting future displacement of nonoperatively managed lateral compression sacral fractures: can it be done? J Orthop Trauma. 2011 Sep;25(9):523-7. doi: 10.1097/BOT.0b013e3181f8be33. PMID 21857419
- [Background] Gaski GE, Manson TT, Castillo RC, Slobogean GP, O'Toole RV. Nonoperative treatment of intermediate severity lateral compression type 1 pelvic ring injuries with minimally displaced complete sacral fracture. J Orthop Trauma. 2014 Dec;28(12):674-80. doi: 10.1097/BOT.0000000000000130. PMID 24740110
- [Background] Kanakaris NK, Angoules AG, Nikolaou VS, Kontakis G, Giannoudis PV. Treatment and outcomes of pelvic malunions and nonunions: a systematic review. Clin Orthop Relat Res. 2009 Aug;467(8):2112-24. doi: 10.1007/s11999-009-0712-2. Epub 2009 Jan 30. PMID 19184260
- [Background] Barei DP, Shafer BL, Beingessner DM, Gardner MJ, Nork SE, Routt ML. The impact of open reduction internal fixation on acute pain management in unstable pelvic ring injuries. J Trauma. 2010 Apr;68(4):949-53. doi: 10.1097/TA.0b013e3181af69be. PMID 19996807
- [Background] Tosounidis T, Kanakaris N, Nikolaou V, Tan B, Giannoudis PV. Assessment of Lateral Compression type 1 pelvic ring injuries by intraoperative manipulation: which fracture pattern is unstable? Int Orthop. 2012 Dec;36(12):2553-8. doi: 10.1007/s00264-012-1685-4. Epub 2012 Oct 25. PMID 23096135
- [Background] Sagi HC, Coniglione FM, Stanford JH. Examination under anesthetic for occult pelvic ring instability. J Orthop Trauma. 2011 Sep;25(9):529-36. doi: 10.1097/BOT.0b013e31822b02ae. PMID 21857421
- [Derived] McKibben NS, O'Hara NN, Slobogean GP, Gaski GE, Nascone JW, Sciadini MF, Natoli RM, McKinley T, Virkus WW, Sorkin AT, Howe A, O'Toole RV, Levy JF. Work Productivity Loss After Minimally Displaced Complete Lateral Compression Pelvis Fractures. J Orthop Trauma. 2024 Jan 1;38(1):42-48. doi: 10.1097/BOT.0000000000002681. PMID 37653607
- [Derived] Slobogean GP, Gaski GE, Nascone J, Sciadini MF, Natoli RM, Manson TT, Lebrun C, McKinley T, Virkus WW, Sorkin AT, Brown K, Howe A, Rudnicki J, Enobun B, O'Hara NN, Gill J, O'Toole RV. A Prospective Clinical Trial Comparing Surgical Fixation Versus Nonoperative Management of Minimally Displaced Complete Lateral Compression Pelvis Fractures. J Orthop Trauma. 2021 Nov 1;35(11):592-598. doi: 10.1097/BOT.0000000000002088. PMID 33993178

RESULTS

PARTICIPANT FLOW:
Groups:
- Operative: Patients enrolled in the operative treatment group will undergo surgical intervention for their pelvic fracture. The surgeon will decide the best surgical technique as per standard of care for the patient's injury. The patient will mobilize as per the surgeon's instructions and x-rays will be taken at follow-up clinic appointments to determine if the injury is healing properly. If additional surgery is required or other complications arise, this will be recorded within the study follow-up forms.
  LC fracture surgical fixation
- Non-operative: Patients enrolled in the non-operative treatment group will not undergo surgical intervention for their pelvic fracture. They will mobilize as per the surgeon's instructions according to standard of care of for this injury. X-rays will be taken at follow-up clinic appointments to determine if the injury is healing properly or if the pelvis has shifted and may warrant surgical intervention. If complications arise and/or surgery is required, crossover will be allowed and recorded within study follow-up forms.
  LC fracture non-operative management
Period: Overall Study
Arm/Group | Operative | Non-operative
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative | Non-operative | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (18.9) | 43.5 (17.9) | 43.5 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 19 | 16 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 46 | 48 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 38 | 39 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Count of Participants; unit: Participants]
  Underweight (< 18.5 kg/m^2) | 2 | 0 | 2
  Normal (18.5-24.9 kg/m^2) | 23 | 29 | 52
  Overweight (25-29.9 kg/m^2) | 15 | 11 | 26
  Obese (>30 kg/m^2) | 7 | 8 | 15
History of Comorbidities [Count of Participants; unit: Participants]
  Comorbidities | 38 | 36 | 74
  No Comorbidities | 9 | 12 | 21
Mechanism of Injury [Count of Participants; unit: Participants]
  Motor Vehicle | 36 | 38 | 74
  Fall | 10 | 9 | 19
  Other | 1 | 1 | 2
Injury Severity Score (ISS) [Mean (Standard Deviation); unit: scores on a scale] — ISS is an internationally recognized scoring system that assesses mortality, morbidity, and other measures of trauma severity. It is based on an anatomical injury severity classification, the Abbreviated Injury Scale (AIS) and is calculated as the sum of the squares of the highest AIS code in each of the three most severely injured ISS body regions. These body regions are: Head or neck, Face, Chest, Abdomen, Extremities (including pelvis), and External.
  ISS ranges from 1 to 75, 1 indicating very few injuries, and 75 indicating virtually unsurvivable injuries.
  scores on a scale | 17 (9) | 18 (10) | 17 (9)
Fracture Type [Count of Participants; unit: Participants] — Lateral compression type 1 (LC1) are defined by an impaction fracture at the sacrum. LC type 2 (LC2) have a fracture that extends through the posterior iliac wing at the level of the sacroiliac joint. Both patterns will have varying amounts of anterior pubic root/rami fractures.
  Participants
    Lateral Compression Type 1 | 31 | 36 | 67
    Lateral Compression Type 2 | 16 | 12 | 28
Initial Fracture Displacement [Count of Participants; unit: Participants]
  <5 mm (no/minimal displacement) | 36 | 33 | 69
  5-10 mm (displaced) | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Posttreatment Pain
Description: The primary outcome was patient-reported pain severity, as measured by the mean of the 4 pain severity items of the Brief Pain Inventory (BPI): worst pain in the last 24 hours, least pain in the last 24 hours, pain on average, and pain right now. The BPI uses a 0-10 level visual analog scale (VAS) with a 24-hour recall period, where 0 anchors "no pain" and 10 anchors "pain as bad as you can imagine." The minimum clinically important difference (MCID) is not definitively established for the BPI in a trauma population; however, the MCID for other 10-point VAS pain scales has been reported between 1.0-2.5 points.
Time Frame: up to 12 weeks post injury
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 47 | 48
scores on a scale
  96 hr | 5.3 (1.8) | 6.2 (2.4)
  2 wk | 4.2 (2.0) | 5.6 (2.3)
  6 wk | 2.7 (2.6) | 3.5 (3.1)
  12 wk | 1.9 (2.0) | 2.9 (2.7)

2. Secondary Outcome: Posttreatment Function
Description: Secondary functional outcome was measured by the Majeed pelvic score. The Majeed pelvic score is a seven-item patient-reported outcome instrument that measures pain, work status, sitting comfort, sexual intercourse, use of walking aids, gait disturbance, and walking distance. The score is reported as a percentage of the highest possible score to adjust for participants who were not employed before their injury. Higher scores represent better function, and a score of >85% has been suggested to represent excellent function.
Time Frame: up to 12 weeks post injury
Measure: Mean (Standard Deviation); unit: percentage of score on a scale
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 47 | 48
percentage of score on a scale
  2 wk | 38 (11) | 31 (10)
  6 wk | 55 (18) | 50 (18)
  12 wk | 73 (20) | 62 (22)

3. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization is determined by recording the admission date versus discharge date for the patient's index hospitalization stay.
Time Frame: through patient discharge, up to 12 weeks post injury
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 47 | 48
days | 6.9 [3.6 to 12.2] | 6.6 [3.4 to 12.4]

4. Secondary Outcome: Time to First Mobilization Post Injury
Description: Time to first mobilization (bed to chair) is determined using the physical therapy notes during the patient's index hospitalization and is recorded as the number of days post injury that mobilization first occurred.
Time Frame: through patient discharge, up to 12 weeks post injury
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Operative | Non-operative
Number analyzed (Participants) | 47 | 48
days | 3 [2 to 5] | 3 [2 to 4.3]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Operative | Non-operative
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 3/47 | 4/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative (N=47) | Non-operative (N=48)
hardware loosening (Surgical and medical procedures) | 2 (2) | 0 (0) — Reoperation due to hardware loosening
Wound seroma requiring drainage (Surgical and medical procedures) | 1 (1) | 0 (0) — Wound seroma requiring drainage
Unplanned fixation (Surgical and medical procedures) | 0 (0) | 4 (4) — Patient randomized to non-operative treatment who later required fixation.

LIMITATIONS AND CAVEATS:
The limitations of the trial are primarily related to its sample size and challenges with recruitment into a randomized controlled trial. The decision to enroll patients who refused randomization, but selected their treatment without surgeon's recommendation, was a study design decision carefully made to balance potential risks of bias with the benefits of increased study power from a larger sample size. Additionally, we acknowledge that we were unable to obtain preoperative pain scores.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02625766/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT02625766/SAP_001.pdf